CLINICAL TRIAL: NCT07001228
Title: Diagnosis and Treatment of Scapular Dyskinesis Combined With Impingement Syndrome of Shoulder
Brief Title: Scapular Dyskinesis With Impingement Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Jung-Taek Hwang, Professor, Chuncheon Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2025-03-009-002
Record Dates: First submitted 2025-05-23; First posted 2025-06-03 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Scapular Dyskinesis; Impingement Syndrome, Shoulder
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Intervention Model Description: This study involves patients who visited the outpatient clinic with unilateral shoulder pain persisting for more than three months and were diagnosed with unilateral shoulder impingement syndrome based on MRI findings. Only patients who provided informed consent were enrolled in the study.
  A total of 320 patients with unilateral shoulder impingement syndrome from Chuncheon Sacred Heart Hospital were included. The participants were randomly assigned into two groups of 160 patients each. Both groups underwent rehabilitation for shoulder impingement syndrome; however, the control group (Group 1) did not receive rehabilitation for scapular dyskinesis, while the experimental group (Group 2) did receive rehabilitation targeting scapular dyskinesis.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The investigators plan to enroll patients who consent to participate in the study and allocate them into two groups using a random sequence generator. A random allocation table will be created and managed by a third party who is not involved in the study. When planning the treatment method, group assignment will be requested from this third party holding the allocation table, ensuring that the allocator is blinded to the upcoming group assignments in advance. Treatment in each group will be administered consistently according to a pre-agreed protocol, and follow-up will also be conducted using the same method in both groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Impinge c SD treatment (Experimental): In this experimental group, rehabilitation for scapular dyskinesis will begin at the second outpatient visit, which takes place three weeks after the subacromial steroid injection.
  Interventions: Behavioral: SD rehabilitation
- Impinge s SD treatment (Sham Comparator): In this sham group, rehabilitation for scapular dyskinesis will not be begun at the second outpatient visit, which takes place three weeks after the subacromial steroid injection.
  Interventions: Behavioral: No SD rehabilitation

INTERVENTIONS:
Behavioral: SD rehabilitation — For shoulder impingement syndrome, the standard rehabilitation protocol involves administering a subacromial steroid injection at the initial outpatient visit, followed by stick exercises to restore joint mobility starting three weeks later. Four weeks after initiating the stick exercises, rotator cuff strengthening exercises using therabands are introduced and maintained for a duration of six weeks.
  For SD rehabilitation, shoulder external rotation, push up plus, and shoulder rolls were performed. In the experimental group, rehabilitation for scapular dyskinesis will begin at the second outpatient visit, which takes place three weeks after the subacromial steroid injection.
  Arms: Impinge c SD treatment
Behavioral: No SD rehabilitation — For shoulder impingement syndrome, the standard rehabilitation protocol involves administering a subacromial steroid injection at the initial outpatient visit, followed by stick exercises to restore joint mobility starting three weeks later. Four weeks after initiating the stick exercises, rotator cuff strengthening exercises using therabands are introduced and maintained for a duration of six weeks.
  In the sham group, rehabilitation for scapular dyskinesis will not begun at the second outpatient visit, which takes place three weeks after the subacromial steroid injection.
  Arms: Impinge s SD treatment

SUMMARY:
The goal of this study is to diagnose scapular dyskinesis-which can appear as a cause or result of various shoulder disorders-through screening tests in patients with shoulder impingement syndrome, the most common shoulder condition. By identifying scapular dyskinesis, the study aims to maximize treatment outcomes through appropriate rehabilitative exercise therapy.

ELIGIBILITY:
1. Inclusion Criteria

   Patients diagnosed with unilateral shoulder impingement syndrome in the outpatient clinic (based on clinical symptoms and MRI) from the IRB approval date until March 1, 2027

   Individuals who provided written informed consent after receiving a thorough explanation of the study prior to any procedures

   Age 20 years or older
2. Exclusion Criteria

Individuals who did not receive a subacromial steroid injection for shoulder impingement syndrome

Individuals with a history of surgical treatment or fracture in the affected shoulder

Individuals who refused to participate in the study

Individuals with neurological disorders affecting the ipsilateral upper extremity

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-05-29 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
visual analog pain scale (VAS) | Initial, 3, 7, 13 weeks
  0-10, 0: not satisfied, 10: very much satisfied

SECONDARY OUTCOMES:
American Shoulder and Elbow Surgeons' (ASES) score | Initial, 3, 7,13 weeks
  0-100
Constant score | Initial, 3, 7, 13 weeks
  0-100

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Taek Hwang, MD, PhD, Principal Investigator — Hallym University Medical Center
Locations (1):
- Hallym University Chuncheon Sacred Heart Hospital, Chuncheon, Gangwon-do, South Korea

IPD SHARING:
Plan to Share IPD: No
We can decide it after the termination of this study.

REFERENCES:
- [Background] Park JY, Hwang JT, Oh KS, Kim SJ, Kim NR, Cha MJ. Revisit to scapular dyskinesis: three-dimensional wing computed tomography in prone position. J Shoulder Elbow Surg. 2014 Jun;23(6):821-8. doi: 10.1016/j.jse.2013.08.016. Epub 2013 Nov 23. PMID 24280352
- [Background] Park JY, Hwang JT, Kim KM, Makkar D, Moon SG, Han KJ. How to assess scapular dyskinesis precisely: 3-dimensional wing computer tomography--a new diagnostic modality. J Shoulder Elbow Surg. 2013 Aug;22(8):1084-91. doi: 10.1016/j.jse.2012.10.046. Epub 2013 Jan 24. PMID 23352185
- [Background] Kibler WB, McMullen J. Scapular dyskinesis and its relation to shoulder pain. J Am Acad Orthop Surg. 2003 Mar-Apr;11(2):142-51. doi: 10.5435/00124635-200303000-00008. PMID 12670140
- [Background] Kibler WB, Ludewig PM, McClure P, Uhl TL, Sciascia A. Scapular Summit 2009: introduction. July 16, 2009, Lexington, Kentucky. J Orthop Sports Phys Ther. 2009 Nov;39(11):A1-A13. doi: 10.2519/jospt.2009.0303. PMID 19881011